CLINICAL TRIAL: NCT07187310
Title: The Analgesic Efficacy of EXORA Block Versus Erector Spinae Plane Block in Patients Undergoing Laparoscopic Cholecystectomy Under General Anesthesia
Brief Title: EXORA vs ESP Blocks in Laparoscopic Cholecystectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Hamed, Professor of Anesthesiology, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: M829
Record Dates: First submitted 2025-09-18; First posted 2025-09-22 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Pain
Keywords: EXORA block; Erector spinae Plain block; Regional Anesthesia for Laparoscopic Cholecystectomy; Postoperative pain management in abdominal surgeries
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EXORA block group (Experimental): Group A (EXORA Block Group): Patients will receive bilateral EXORA blocks.
  Interventions: Procedure: EXORA block
- ESP block group (Active Comparator): Group B (ESP Block Group): Patients will receive bilateral ESP blocks.
  Interventions: Procedure: Erector Spinae Plane block
- control group (No Intervention): Group C (Control Group): patients will not receive any block, only standard care.

INTERVENTIONS:
Procedure: EXORA block — in a supine position, a linear Ultrasound probe (L6-12 RS linear array transducer (6-12 MHz) on GE Healthcare Logiq P7, made in Korea) will be sagittally applied at the parasternal line, lateral to the sternum and xiphoid process. The probe will be manipulated craniocaudally to identify the 6th, 7th, and 8th costal cartilages. At the level of the 8th costal cartilage, a transverse orientation will be used to visualize the rectus abdominis muscle and the costal cartilage beneath. An 88-mm, 22-gauge needle will be directed in-plane from medial to lateral. After confirming the needle position below the rectus abdominis muscle using 4 ml isotonic saline as a hydro-dissection, 25 ml of plain bupivacaine 0.25% concentration will be injected. the spread of the local anesthetic is to be observed to advance laterally under the external oblique muscle and medially under the rectus muscle. The same procedure will be repeated on the other side.
  Arms: EXORA block group
Procedure: Erector Spinae Plane block — in a right lateral position, the linear Ultrasound probe will be placed vertically 3 cm lateral to the midline at the level of the 7th thoracic spinal process, identifying the T7 transverse process, and the overlying erector spinae (ES) muscle. An 88-mm, 22-gauge needle will be advanced craniocaudally in-plane until hitting the T7 transverse process. After using hydro-dissection with 4 ml of isotonic saline to confirm the correct needle position, 25 ml of 0.25% bupivacaine will be administered below the erector spinae muscle. The same procedure will be repeated on the other side.
  Arms: ESP block group

SUMMARY:
Laparoscopic cholecystectomy is still considered the gold standard for the surgical management of gallbladder disease due to its minimally invasive nature, shorter recovery time, and reduced postoperative complications. Despite these advantages, patients frequently experience moderate to severe postoperative pain, particularly in the early postoperative period, which can impede recovery, delay mobilization, and increase opioid consumption. Excessive opioid use after laparoscopic cholecystectomy is associated with several drawbacks, including nausea, vomiting, sedation, and delayed recovery. It also increases the risk of respiratory depression, especially in vulnerable patients, and may contribute to long-term opioid dependence. These risks highlight the importance of opioid-sparing strategies such as regional anesthesia techniques to improve patient outcomes and enhance recovery. Regional anesthesia techniques have emerged as essential components of multimodal analgesia strategies in abdominal surgeries. Among them, the Erector Spinae Plane (ESP) Block has gained popularity due to its relative ease of administration and favorable safety profile.

Recently, a novel fascial plane block known as the EXORA block has been introduced as a promising alternative for abdominal wall analgesia. This block, which targets a different anatomical plane, is postulated to provide comparable or superior analgesic efficacy to traditional methods while maintaining safety and simplicity in execution. Given the ongoing pursuit of optimal analgesia with minimal side effects, it is essential to compare emerging techniques, such as the EXORA block, with established methods like the ESP block.

The authors hypothesize that the EXORA and the ESP blocks provide superior postoperative analgesia compared to controls in the anterolateral abdomen in patients undergoing laparoscopic cholecystectomy and that the EXORA block analgesic profile is comparable to that of the ESP block.

DETAILED DESCRIPTION:
Following the tenets of the Declaration of Helsinki and the Consolidated Standards of Reporting Trials (CONSORT) 2025-updated statement, this prospective, randomized, double-blinded, controlled clinical trial will be conducted at Fayoum University Hospital (FUH) starting from October 2025 until the sample size is reached.

After obtaining approval from the local institutional ethics committee at Fayoum University Hospital (FUH) and registering the trial on ClinicalTrials.gov, all patients scheduled for elective cholecystectomy at FUH will sign a detailed informed consent form after fulfilling the eligibility criteria.

Patients will be randomly assigned to three equal groups with an allocation ratio of 1:1:1 (n=35) using computer-generated random numbers that will be sealed in a closed opaque envelope, opened by the anesthesiologist responsible for administering the ultrasound-guided block preoperatively

* Group A (EXORA Block Group): Patients will receive bilateral EXORA blocks.
* Group B (ESP Block Group): Patients will receive bilateral ESP blocks.
* Group C (Control Group): patients will not receive any block, only standard care.

Preoperatively, all patients will be assessed and investigated by complete blood count, Prothrombin time and concentration, kidney and liver functions. Additional investigations, such as serum electrolytes, ECG, ECHO, etc., will be ordered upon individual patient assessment.

All blocks will be performed by an anesthesiologist experienced in regional blocks preoperatively in a separate block room under strict aseptic conditions using ultrasound guidance after applying standard monitoring (pulse oximetry, non-invasive blood pressure, and electrocardiogram) and administering a sedative dose of intravenous midazolam (0.03 mg/kg).

For both groups A and B, sensory block will be assessed by a blinded anesthesiologist after 30 minutes from the block maneuver bilaterally from the distribution of the fifth Thoracic dermatome (T5) down to the level of the twelfth thoracic dermatome (T12). This will be accomplished using a pinprick with a blunt 20-G needle on a two-point scale, where 0 indicates the presence of sensation and 1 indicates numbness or absence of sensation in reference to sensation in the shoulder region. If no sensory loss is observed, the patient will be excluded from the study.

All patients will then be transferred to the operating room, handed over to the attending anesthesiologist who is blinded to group allocation and is responsible for further patient management. standard monitoring will be reapplied, and then general anesthesia will be induced using propofol (2 mg/kg), atracurium (0.5 mg/kg), and fentanyl (2 μg/kg). Anesthesia will be maintained with intermittent intravenous atracurium (0.1 mg/kg boluses) and an isoflurane inhalation in an oxygen and air mixture. An intravenous Ketorolac (30 mg), Nalbuphine (10 mg), and Ondansetron 8 mg will be administered approximately 30 minutes before the end of the operation.

After discharge to the ward, paracetamol 1g /8 hours and ketorolac 30 mg/12 hours will be administered to all patients. Both static (at rest) and dynamic (with movement) visual analogue scale (VAS) will be assessed at 1,2, 4, 6, 12, and 24 hours (where 0 denotes no pain, and 10 represents the most intense pain ever experienced), and if the VAS score is equal to or higher than 4, a rescue analgesic dose of nalbuphine 5 mg will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Elective laparoscopic cholecystectomy
* ASA physical status I-III

Exclusion Criteria:

* Known allergy to local anesthetics
* Chronic pain or regular opioid use
* Coagulopathy or anticoagulant therapy
* Local infection at the block site
* BMI more than 35 kg/m2
* Neurological or psychiatric disorders
* Refusal to participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2025-12-30 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Total opioid consumption | Up to 24 hours after surgery
  Post operative nalbuphine used in the first 24 hours in milligrams

SECONDARY OUTCOMES:
Intraoperative Fentanyl consumption | From induction of anesthesia until patient is transferred to postoperative care unit up to 4 hours
  Total fentanyl in milligrams
Time needed to complete the block | From start of block procedure up to 1 hour
  In minutes
Sensory block distribution level (pin-prick test) | after 30 minuets from the block maneuver bilaterally
  sensory block will be assessed by a blinded anesthesiologist after 30 minutes from the block maneuver bilaterally from the distribution of the fifth Thoracic dermatome (T5) down to the level of the twelfth thoracic dermatome (T12). This will be accomplished using a pinprick with a blunt 20-G needle on a two-point scale, where 0 indicates the presence of sensation and 1 indicates numbness or absence of sensation in reference to sensation in the shoulder region.
Heart rate | Upon arrival to Operating Room until 24 hours postoperative
  Heart rate (HR) recorded intra and post operative
Blood pressure | Upon arrival to Operating Room until 24 hours postoperative
  Mean Arterial Pressure (MAP)
Postoperative pain scores by Visual Analogue Scale (VAS) | From patient discharge to postoperative anesthesia care unit 24 hours postoperatively
  score from 0 to 10 where 0 indicates no pain and 10 indicates the worst imaginable pain
Rescue analgesia | Upon recovery from General anesthesia up to 24 h postoperatively
  Time to first request of rescue analgesia
Incidence of opioid-related side effects | From induction of anesthesia up to 24 h postoperatively
  Assessment of each patient looking for any of the side effects of opioids as nausea, vomiting, sedation.
Incidence of Block-related side effects | From the time just after giving the block up to 24 h postoperatively
  any Block-related side effects as Local anesthetic systemic toxicity, bleeding, pneumothorax, local infection.

OTHER OUTCOMES:
Quality of recovery (QoR-15) | At 24 hours postoperatively
  scores range from 0 to 150, with a higher score indicating a better quality of postoperative recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Hamed, MD, Principal Investigator — Faculty of medicine, Fayoum university
Locations (1):
- Fayoum University hospital, El Fayoum Qesm, Faiyum Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Asad U, Wang CF, Jones MW. Laparoscopic Cholecystectomy. 2025 Jul 2. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK448145/ PMID 28846328
- [Background] Roy DK, Sheikh R. A Systematic Review and Meta-Analysis of the Outcomes of Laparoscopic Cholecystectomy Compared to the Open Procedure in Patients with Gallbladder Disease. Avicenna J Med. 2024 Feb 1;14(1):3-21. doi: 10.1055/s-0043-1777710. eCollection 2024 Jan. PMID 38694141
- [Background] Ekstein P, Szold A, Sagie B, Werbin N, Klausner JM, Weinbroum AA. Laparoscopic surgery may be associated with severe pain and high analgesia requirements in the immediate postoperative period. Ann Surg. 2006 Jan;243(1):41-6. doi: 10.1097/01.sla.0000193806.81428.6f. PMID 16371735
- [Background] Dua A, Aziz A, Desai SS, McMaster J, Kuy S. National Trends in the Adoption of Laparoscopic Cholecystectomy over 7 Years in the United States and Impact of Laparoscopic Approaches Stratified by Age. Minim Invasive Surg. 2014;2014:635461. doi: 10.1155/2014/635461. Epub 2014 Mar 20. PMID 24790759
- [Background] Urman RD, Khanna AK, Bergese SD, Buhre W, Wittmann M, Le Guen M, Overdyk FJ, Di Piazza F, Saager L. Postoperative opioid administration characteristics associated with opioid-induced respiratory depression: Results from the PRODIGY trial. J Clin Anesth. 2021 Jun;70:110167. doi: 10.1016/j.jclinane.2021.110167. Epub 2021 Jan 22. PMID 33493688
- [Background] Lohmoller K, Carstensen V, Pogatzki-Zahn EM, Freys SM, Weibel S, Schnabel A. Regional anaesthesia for postoperative pain management following laparoscopic, visceral, non-oncological surgery a systematic review and meta-analysis. Surg Endosc. 2024 Apr;38(4):1844-1866. doi: 10.1007/s00464-023-10667-w. Epub 2024 Feb 2. PMID 38307961
- [Background] Sethi D, Garg G. Evaluation of postoperative analgesia of erector spinae plane block in elective laparoscopic cholecystectomy: a randomized controlled trial. Turk J Anaesthesiol Reanim. 2021 Dec;49(6):432-438. doi: 10.5152/TJAR.2021.878. PMID 35110021
- [Background] Altiparmak B, Korkmaz Toker M, Uysal AI, Kuscu Y, Gumus Demirbilek S. Ultrasound-guided erector spinae plane block versus oblique subcostal transversus abdominis plane block for postoperative analgesia of adult patients undergoing laparoscopic cholecystectomy: Randomized, controlled trial. J Clin Anesth. 2019 Nov;57:31-36. doi: 10.1016/j.jclinane.2019.03.012. Epub 2019 Mar 6. PMID 30851501
- [Background] Yang X, Zhang Y, Chen Y, Xu M, Lei X, Fu Q. Analgesic effect of erector spinae plane block in adults undergoing laparoscopic cholecystectomy: a systematic review and meta-analysis of randomized controlled trials. BMC Anesthesiol. 2023 Jan 6;23(1):7. doi: 10.1186/s12871-023-01969-6. PMID 36609244
- [Background] Fernandez Martin MT, Lopez Alvarez S, Valdes-Vilches LF. EXORA block: a new approach for laparoscopic cholecystectomy analgesia? Minerva Anestesiol. 2024 May;90(5):462-463. doi: 10.23736/S0375-9393.23.17863-1. Epub 2024 Jan 29. No abstract available. PMID 38287777
- [Background] Okmen K, Yildiz DK, Ulker GK. Evaluation of the efficacy of M-TAPA and EXORA block application for analgesia after laparoscopic cholecystectomy: a prospective, single-blind, observational study. Korean J Anesthesiol. 2025 Aug;78(4):361-368. doi: 10.4097/kja.24563. Epub 2025 Apr 15. PMID 40230270